CLINICAL TRIAL: NCT03094611
Title: Phase II Study of Low Dose Inotuzumab Ozogamicin in Patients With Relapsed and Refractory CD22 Positive Acute Lymphocytic Leukemia
Brief Title: Inotuzumab Ozogamicin in Treating Patients With Relapsed or Refractory CD22 Positive Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study was closed early due to competing trials
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0870; NCI-2018-01237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0870 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: CD22 Positive; Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (inotuzumab ozogamicin) (Experimental): Patients receive inotuzumab ozogamicin IV over 1 hour on days 1, 8 and 15 of cycle 1 and on days 1 and 8 beginning cycle 2. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients whose disease gets worse after responding for 3 months, may be retreated for up to 6 additional cycles. Patients whose disease responds to treatment may receive up to 5 additional cycles.
  Interventions: Biological: Inotuzumab Ozogamicin

INTERVENTIONS:
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294

SUMMARY:
This phase II trial studies how well inotuzumab ozogamicin works in treating patients with CD22 positive acute lymphoblastic leukemia that has come back or does not respond to treatment. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called ozogamicin. Inotuzumab attaches to CD22 positive cancer cells in a targeted way and delivers ozogamicin to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate of low dose of inotuzumab ozogamicin as measured by the hematologic remission rate (complete remission [CR] + CR with incomplete platelet recovery [CRp] + CR with incomplete bone marrow recovery [CRi]) in patients in first, second or later salvage setting.

SECONDARY OBJECTIVES:

I. To evaluate the overall safety profile and the efficacy; the efficacy is measured by the hematologic response rate (CR + CRi + PR), durations of response (DoR) and remission (DoR1), progression free survival (PFS), and overall survival (OS).

OUTLINE:

Patients receive inotuzumab ozogamicin intravenously (IV) over 1 hour on days 1, 8 and 15 of cycle 1 and on days 1 and 8 beginning cycle 2. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients whose disease gets worse after responding for 3 months, may be retreated for up to 6 additional cycles. Patients whose disease responds to treatment may receive up to 5 additional cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 12 years of age
* Patients with a diagnosis of CD22-positive acute lymphoblastic leukemia (ALL) based on local immunophenotyping and histopathology who have:

  * Refractory disease, defined as disease progression or no response while receiving their most recent prior anti-cancer therapy,
  * Relapsed disease, defined as response to their most recent prior anti-cancer therapy with subsequent relapse
* Performance status of 0 to 3
* Serum creatinine =< 2 x upper limit of normal (ULN) or estimated creatinine clearance >= 15 mL/min as calculated using the method standard for the institution
* Total serum bilirubin =< 1.5 x ULN unless the patient has documented Gilbert syndrome. If organ function abnormalities are considered due to tumor, total serum bilirubin must be =< 2 x ULN
* Aspartate and alanine aminotransferase (AST or ALT) =< 2.5 x ULN
* No active or co-existing malignancy requiring chemotherapy or radiation within 6 months
* Female subjects of childbearing potential should be willing to use effective methods birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Effective methods of birth control include birth control pills or injections, intrauterine devices (IUDs), or double-barrier methods (for example, a condom in combination with spermicide)
* Male subjects should agree to use an effective method of contraception starting with the first dose of study therapy through the duration of treatment

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus (HIV)+
* Philadelphia chromosome (Ph)+ ALL
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Prior allogeneic stem cell transplantation (ASCT) or other anti-CD22 immunotherapy within =< 4 months before first dose of study treatment
* Active central nervous system (CNS) or extramedullary disease unless approved by the principal investigator (PI)
* Monoclonal antibodies therapy within 2 weeks before study entry
* Radiotherapy and cancer chemotherapy (except for intrathecal chemotherapy, hydroxyurea, and cytarabine. Cytarabine and hydroxyurea are allowed to be used emergently in case of leukocytosis) or any investigational drug within 2 weeks before study entry
* Evidence or history of veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2017 to January 2019
Period: Overall Study
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Started | 4
Completed | 2
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Stem Cell Transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 46 [32 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Achieve Complete Remission (CR)
Description: Complete Remission (CR) is the normalization of the peripheral blood and bone marrow with </= 5% blasts with a granulocyte count of 1X10^9/L or above and a platelet count of >/= 100X10^9/L and absence of extramedullary disease.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Participants | 3

2. Secondary Outcome: Participants With a Grade 3 or 4 Non-hematologic Adverse Event (AE)
Description: For the purpose of toxicity monitoring, toxicities are defined as any treatment -related grade 3 or 4 non-hematologic AEs occurred any time during the trial.NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 utilized for adverse event reporting.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Participants | 1

3. Secondary Outcome: Duration of Response
Description: The date of Complete Response to the date of loss of response or last follow-up.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Months | 17.0 [11.1 to 31.8]

4. Secondary Outcome: Progression Free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Months | 11.7 [0.4 to 32.7]

5. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Months | 19.6 [1.5 to 32.7]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Inotuzumab Ozogamicin)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Inotuzumab Ozogamicin) (N=4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Inotuzumab Ozogamicin) (N=4)
Alkaline Phosphatase Increased (Investigations) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 3 (3)
Hyperbilirubinemia (Investigations) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine Aminotransferase Increase (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03094611/Prot_SAP_000.pdf